CLINICAL TRIAL: NCT02747121
Title: Effects of External Inspection on Sepsis Detection and Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Board of Health Supervision (Other Government)
Collaborators: University of Bergen (Other); Norwegian Institute of Public Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 2015/2195 REK number
Record Dates: First submitted 2016-04-11; First posted 2016-04-21 (Estimated); Results first posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-01

CONDITIONS: Sepsis
Keywords: External inspections
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Intervention Model Description: The intervention will be rolled out sequentially during 12 months to 24 hospitals, with six clusters of four geographically close hospitals. We collect data before and after the inspections.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control before intervention (Other): External inspection of health services. The intervention is external inspection of sepsis detection and treatment. The intervention is delivered on the organizational Level. Patient are not assigned to the intervention. The intervention is rolled out sequentially to 24 hospitals. We collect data at base line, before the inspections and 8 and 14 month after the inspections. The first arm is the Control period before the inspections.
  Interventions: Behavioral: External inspection of health services
- Intervention (Experimental): External inspection of health services. We compare the effect measures before and after the inspection. The intervention arm is data after the hospitals have received the inspection.
  Interventions: Behavioral: External inspection of health services

INTERVENTIONS:
Behavioral: External inspection of health services — The intervention is external inspections of acute hospitals addressing early detection and treatment of sepsis. The intervention is delivered on an organizational level. Individuals are not assigned to an intervention. The investigator use data from individuals to assess if the organizational intervention affects care. Therefore the investigator argues that that the study is observational. The inspection will have two components, a system revision and a follow up audit with verification of patient records 8 months later. The inspection can be considered a complex intervention. The study does not intend to evaluate the individual effects of the different components of the inspection, rather the effect of the inspection as a whole.

SUMMARY:
External inspections are widely used as means to improve the quality of care. Despite their widespread use, there is limited knowledge about whether and how they affect the quality of care. This study uses inspection with detection and treatment of sepsis in hospitals as a case to evaluate the effect of inspections on the quality of care and to explore how inspections affect the hospitals.

DETAILED DESCRIPTION:
The aim of this study is to assess what effect external inspections have on the quality of care provided to sepsis patients admitted to hospital and to explore how external inspections affect the involved organizations.

External inspections are widely used as a means to improve the quality of care, and it is a core element of regulatory regimes and certification and accreditation processes. The activity of assessing a health care organization's performance according to an externally defined standard has been described by partly overlapping terms such as external inspection, external review, supervision, and audit. The project uses the term external inspection implying that the inspection is initiated and controlled by an organization external to the one being inspected; and define it as: "a system, process or arrangement in which some dimensions or characteristics of a healthcare provider organisation and its activities are assessed or analysed against a framework of ideas, knowledge, or measures derived or developed outside that organisation".

In line with this definition the investigator intend to study how external inspection affect the quality of care provided on an organizational level. The project does not intend to study how external inspections can affect individuals in the organization nor individual professional development. The investigator takes the perspective that quality of care can be considered a system property, being dependent on how the organization providing care performs as a whole. Accordingly, improving the quality of care is dependent on changing the performance of the organization, which in turn implies change in organizational behavior and the way clinicians mutually interact and perform their clinical processes. Change in organizational behavior is a complex social process that involves a number of different practices on different organizational levels. If external inspection has the ability to contribute to improve the quality of care on an organizational level, it need to affect the practices involved in organizational change.

The effect of external inspection systems on the quality of care remains unclear and the evidence is contradictory. Studies have demonstrated a positive association between accreditation and the ability to promote change, professional development, quality systems, and clinical leadership. There is evidence to support an association between inspections and different quality outcomes e.g. reduced incidence of pressure ulcer and suicide. There are however also studies reporting that inspections have no impact on the quality of care. Inspection systems are widely used and much resources are spent on such systems worldwide. More knowledge about how and whether external inspections can effect the quality of care is needed.

The inspection process can be considered a complex intervention consisting of a set of activities that are introduced into varying organizational contexts. The inspection itself does not have a direct impact on the quality of care. If the inspection encounters non-compliant behavior, the inspected organization is responsible for implementing necessary changes. The way the inspection process affects the involved organization will thus influence how the inspected organizations pursue the following change process. The way external inspections affect the involved organization, is currently poorly understood. A better understanding of the underlying mechanisms for how inspection systems might contribute to improve the quality of care is needed. Such knowledge can improve the understanding of why effects of external inspections seem to vary, which in turn can facilitate the development of more effective ways of conducting inspections.

The study uses external inspections of sepsis detection and treatment in hospitals as a case to explore how inspections affect the involved organizations and to evaluate their effect on the quality of care. Sepsis is a prevalent disease and one of the main causes of death among hospitalized patients internationally and in Norway. Former external inspections of Norwegian hospitals have showed that insufficient governance of clinical process in the emergency room could have severe consequences for patients admitted to hospital with undiagnosed sepsis. During recent years, the Norwegian Board of Health Supervision has investigated a number of cases in which the hospitals had not provided care in line with the recommended guidelines for sepsis treatment. On this background, the Norwegian Board of Health Supervision has decided to conduct a nationwide inspection campaign with sepsis detection and treatment in acute hospitals during 2016-2017.

Early treatment with antibiotics along with compliance to treatment guidelines is associated with reduced mortality for sepsis patients. International studies have shown that compliance with treatment guidelines varies, and that improved compliance can improve patient outcomes. External inspection can identify sub-optimal compliance with treatment guidelines. Improved compliance with treatment guidelines is dependent on change in organizational practice. Such changes in organizational practice can be measured using process indicators that are indicative and sensitive for changes in the key areas identified during the inspection. The study uses process measures to assess how external inspections affect guideline adherence. Because improved guideline adherence has been demonstrated to improve the quality of care in terms of reduced mortality, it can be argued that this is an expedient case for evaluating how external inspections can affect the quality of care.

ELIGIBILITY:
Inclusion Criteria:

* Suspected infection and minimum 2 SIRS criteria. If high leucocytes are one of the two criteria, then 3 SIRS criteria are needed.

Exclusion Criteria:

* Patients below the age of 18 years.
* Patients who do not pass through the emergency room.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7407 (Actual)
Dates: Start 2016-04; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Fredrik Andresen, MD, Study Chair — Head of Norwegian Board of Health Supervision
Locations (1):
- Haukeland hospital, Bergen, Hordaland, Norway

IPD SHARING:
Plan to Share IPD: No
In line with the ethical approval data is not to be shared outside the research group

REFERENCES:
- [Background] Walshe K, Wallace L, Freeman T, Latham L, Spurgeon P. The external review of quality improvement in health care organizations: a qualitative study. Int J Qual Health Care. 2001 Oct;13(5):367-74. doi: 10.1093/intqhc/13.5.367. PMID 11669564
- [Background] van Dishoeck AM, Oude Wesselink SF, Lingsma HF, Steyerberg E, Robben PB, Mackenbach JP. [Transparency: can the effect of governmental surveillance be quantified?]. Ned Tijdschr Geneeskd. 2013;157(16):A1676. Dutch. PMID 23594866
- [Background] Shaw CD, Braithwaite J, Moldovan M, Nicklin W, Grgic I, Fortune T, Whittaker S. Profiling health-care accreditation organizations: an international survey. Int J Qual Health Care. 2013 Jul;25(3):222-31. doi: 10.1093/intqhc/mzt011. Epub 2013 Feb 13. PMID 23411832
- [Background] Oude Wesselink SF, Lingsma HF, Reulings PG, Wentzel HR, Erasmus V, Robben PB, Mackenbach JP. Does government supervision improve stop-smoking counseling in midwifery practices? Nicotine Tob Res. 2015 May;17(5):572-9. doi: 10.1093/ntr/ntu190. Epub 2014 Sep 19. PMID 25239965
- [Background] Plsek PE, Greenhalgh T. Complexity science: The challenge of complexity in health care. BMJ. 2001 Sep 15;323(7313):625-8. doi: 10.1136/bmj.323.7313.625. No abstract available. PMID 11557716
- [Background] Miller RR 3rd, Dong L, Nelson NC, Brown SM, Kuttler KG, Probst DR, Allen TL, Clemmer TP; Intermountain Healthcare Intensive Medicine Clinical Program. Multicenter implementation of a severe sepsis and septic shock treatment bundle. Am J Respir Crit Care Med. 2013 Jul 1;188(1):77-82. doi: 10.1164/rccm.201212-2199OC. PMID 23631750
- [Background] Levy MM, Rhodes A, Phillips GS, Townsend SR, Schorr CA, Beale R, Osborn T, Lemeshow S, Chiche JD, Artigas A, Dellinger RP. Surviving Sepsis Campaign: association between performance metrics and outcomes in a 7.5-year study. Crit Care Med. 2015 Jan;43(1):3-12. doi: 10.1097/CCM.0000000000000723. PMID 25275252
- [Background] Levy MM, Dellinger RP, Townsend SR, Linde-Zwirble WT, Marshall JC, Bion J, Schorr C, Artigas A, Ramsay G, Beale R, Parker MM, Gerlach H, Reinhart K, Silva E, Harvey M, Regan S, Angus DC; Surviving Sepsis Campaign. The Surviving Sepsis Campaign: results of an international guideline-based performance improvement program targeting severe sepsis. Crit Care Med. 2010 Feb;38(2):367-74. doi: 10.1097/CCM.0b013e3181cb0cdc. PMID 20035219
- [Background] Institute of Medicine (US) Committee on Quality of Health Care in America. Crossing the Quality Chasm: A New Health System for the 21st Century. Washington (DC): National Academies Press (US); 2001. Available from http://www.ncbi.nlm.nih.gov/books/NBK222274/ PMID 25057539
- [Background] Gatewood MO, Wemple M, Greco S, Kritek PA, Durvasula R. A quality improvement project to improve early sepsis care in the emergency department. BMJ Qual Saf. 2015 Dec;24(12):787-95. doi: 10.1136/bmjqs-2014-003552. Epub 2015 Aug 6. PMID 26251506
- [Background] Flodgren G, Pomey MP, Taber SA, Eccles MP. Effectiveness of external inspection of compliance with standards in improving healthcare organisation behaviour, healthcare professional behaviour or patient outcomes. Cochrane Database Syst Rev. 2011 Nov 9;(11):CD008992. doi: 10.1002/14651858.CD008992.pub2. PMID 22071861
- [Background] Flaatten H. Epidemiology of sepsis in Norway in 1999. Crit Care. 2004 Aug;8(4):R180-4. doi: 10.1186/cc2867. Epub 2004 May 14. PMID 15312216
- [Background] Ferrer R, Artigas A, Levy MM, Blanco J, Gonzalez-Diaz G, Garnacho-Montero J, Ibanez J, Palencia E, Quintana M, de la Torre-Prados MV; Edusepsis Study Group. Improvement in process of care and outcome after a multicenter severe sepsis educational program in Spain. JAMA. 2008 May 21;299(19):2294-303. doi: 10.1001/jama.299.19.2294. PMID 18492971
- [Background] Campbell M, Fitzpatrick R, Haines A, Kinmonth AL, Sandercock P, Spiegelhalter D, Tyrer P. Framework for design and evaluation of complex interventions to improve health. BMJ. 2000 Sep 16;321(7262):694-6. doi: 10.1136/bmj.321.7262.694. No abstract available. PMID 10987780
- [Background] Donabedian A. The quality of care. How can it be assessed? JAMA. 1988 Sep 23-30;260(12):1743-8. doi: 10.1001/jama.260.12.1743. PMID 3045356
- [Background] Brubakk K, Vist GE, Bukholm G, Barach P, Tjomsland O. A systematic review of hospital accreditation: the challenges of measuring complex intervention effects. BMC Health Serv Res. 2015 Jul 23;15:280. doi: 10.1186/s12913-015-0933-x. PMID 26202068
- [Background] Berwick DM. Crossing the boundary: changing mental models in the service of improvement. Int J Qual Health Care. 1998 Oct;10(5):435-41. doi: 10.1093/intqhc/10.5.435. PMID 9828033
- [Background] Barochia AV, Cui X, Vitberg D, Suffredini AF, O'Grady NP, Banks SM, Minneci P, Kern SJ, Danner RL, Natanson C, Eichacker PQ. Bundled care for septic shock: an analysis of clinical trials. Crit Care Med. 2010 Feb;38(2):668-78. doi: 10.1097/CCM.0b013e3181cb0ddf. PMID 20029343
- [Background] Angus DC, Linde-Zwirble WT, Lidicker J, Clermont G, Carcillo J, Pinsky MR. Epidemiology of severe sepsis in the United States: analysis of incidence, outcome, and associated costs of care. Crit Care Med. 2001 Jul;29(7):1303-10. doi: 10.1097/00003246-200107000-00002. PMID 11445675
- [Derived] Husabo G, Nilsen RM, Solligard E, Flaatten HK, Walshe K, Frich JC, Bondevik GT, Braut GS, Helgeland J, Harthug S, Hovlid E. Effects of external inspections on sepsis detection and treatment: a stepped-wedge study with cluster-level randomisation. BMJ Open. 2020 Oct 20;10(10):e037715. doi: 10.1136/bmjopen-2020-037715. PMID 33082187
- [Derived] Hovlid E, Frich JC, Walshe K, Nilsen RM, Flaatten HK, Braut GS, Helgeland J, Teig IL, Harthug S. Effects of external inspection on sepsis detection and treatment: a study protocol for a quasiexperimental study with a stepped-wedge design. BMJ Open. 2017 Sep 5;7(9):e016213. doi: 10.1136/bmjopen-2017-016213. PMID 28877944

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control Before Intervention
Started | 3594 | 3813
Completed | 3594 | 3813
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: As this was stepped wedge trial we used the pre-intervention measurements as baseline (control group)
Groups:
- After Intervention (After Inspection): Patients included after intervention.
  External inspection of health services: The intervention is external inspections of acute hospitals addressing early detection and treatment of sepsis. The intervention is delivered on an organizational level. Individuals are not assigned to an intervention. The investigator use data from individuals to assess if the organizational intervention affects care. Therefore the investigator argues that that the study is observational. The inspection will have two components, a system revision and a follow up audit with verification of patient records 8 months later. The inspection can be considered a complex intervention. The study does not intend to evaluate the individual effects of the different components of the inspection, rather the effect of the inspection as a whole.
- Total: Total of all reporting groups
Arm/Group | Control Before Intervention | After Intervention (After Inspection) | Total
Number analyzed (Participants) | 3813 | 3594 | 7407
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 70 [56 to 81] | 73 [60 to 82] | 72 [58 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1874 | 1713 | 3587
  Male | 1939 | 1881 | 3820
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Sepsis Patients With 30 Days Mortality
Description: We will still use 30-day mortality rate as our outcome measure. The new international sepsis definition will over time affect coding practice and we can therefore not use routine data from the National Patient Register to calculate the mortality rate. We will calculate the mortality rate based on the patient population we include in the study. We will compare mortality rates before and after the inspections.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control Before Intervention
Number analyzed (Participants) | 3594 | 3813
Participants
  Decesed Deceased within 30 days | 377 | 424
  Alive within 30 days | 3217 | 3389
Statistical Analysis 1: Comparison: Control Before Intervention; Test type: Other — The intervention was external inspections. This is an organizational level intervention and it does not replace any existing intervention; p = 0.24, Mixed Models Analysis — We used calculated P-values, however only confidence intervals were reported in the published article; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.86 to 1.80]

2. Secondary Outcome: Hospital Length of Stay
Description: Mean time for hospital length of stay before and after inspections
Time Frame: Exact number of days for the length of stay was collected from the National Patient Registry. Since the outcome measure is length of stay, the time frame varies between patients. Time frame for observation periode was at least 12 months for each patient.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention | Control Before Intervention
Number analyzed (Participants) | 3594 | 3813
days | 6.2 (6.1) | 7.1 (7.8)

ADVERSE EVENTS:
Time Frame: Intervention was delivered on the organizational level and not to individuals, thus we did not monitor adverse events.
Description: The study did not monitor adverse events
Arm/Group | Intervention | Control Before Intervention
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/21/NCT02747121/Prot_SAP_000.pdf